CLINICAL TRIAL: NCT06634745
Title: Evaluation of the Effectiveness of Antimicrobial Photodynamic Therapy Using Different Irrigation Activation Techniques in Teeth With Apical Periodontitis: A Randomized Controlled Clinical Trial
Brief Title: The Effect of Antimicrobial Photodynamic Therapy on the Success of Root Canal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/058
Record Dates: First submitted 2024-09-27; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2023-05

CONDITIONS: Antimicrobial Photodynamic Therapy
Keywords: Antimicrobial photodynamic therapy; Methylene blue; Apical periodontitis
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Intervention Model Description: This study is a randomized, parallel-group clinical trial evaluating the effectiveness of antimicrobial photodynamic therapy (aPDT) using different irrigation activation techniques in teeth with apical periodontitis. Sixty patients with single-rooted, single-canal teeth were included. Participants were randomly assigned to four groups: aPDT with standard needle irrigation (SII), aPDT with Endoactivator, aPDT with passive ultrasonic irrigation (PUI), and aPDT with EDDY. All groups received aPDT using methylene blue, following standard endodontic procedures. The primary outcome was the efficacy of microbial reduction in the root canal system. Secondary outcomes included lesion healing, postoperative pain, and discoloration potential. Data were analyzed to compare the effectiveness of different techniques. The null hypothesis was that there would be no significant difference among the groups in terms of lesion healing, postoperative pain, and discoloration potential.
Who Masked: Participant
Masking Description: Participants: The participants in this study were blinded to their treatment allocation. They did not know whether they were receiving antimicrobial photodynamic therapy (aPDT) with standard needle irrigation, EDDY sonic activation system, passive ultrasonic irrigation, or Endoactivator sonic activation system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard Needle Irrigation (SNI) with MB Activation (Experimental): In this group, the activation of MB (Merck KgaA) was performed using a 30G NaviTip (Cermaked) with 1 activation cycle. The 30G NaviTip (Cermaked) was placed in the root canal 1 mm short of the working length and used with a 3-4 mm amplitude. The MB (Merck KgaA) solution was activated for 1 minute and renewed during the treatment
  Interventions: Procedure: Standard Needle Irrigation (SNI)
- Passive Ultrasonic Irrigation (PUI) with MB Activation (Experimental): In this group, the activation of MB (Merck KgaA) was performed using Ultra X (Eighteeth, Changzhou, China) and a #25 ultrasonic endodontic tip (Eighteeth) at a frequency of 45 kHz. The ultrasonic endodontic tip was placed in the root canal 1 mm short of the working length and the MB (Merck KgaA) solution was activated for 1 minute. During the activation process, care was taken to ensure the ultrasonic endodontic tip moved freely within the canal, and the MB solution was renewed during the treatment.
  Interventions: Procedure: Passive Ultrasonic Irrigation (PUI
- EndoActivator(EA) with MB Activation (Experimental): In this group, the activation of MB (Merck KgaA) was performed using a polymer EA tip (Dentsply, Tulsa, OK) with a 25.04 tip diameter, which was placed into the canal 2 mm short of the working length. The activation procedure was carried out for 1 minute using the EA sonic irrigation device at 10,000 cycles, and the MB (Merck KgaA) solution was renewed during the treatment.
  Interventions: Procedure: EndoActivator (EA)
- EDDY with MB Activation (Experimental): In this group, the activation of MB (Merck KgaA) was performed using a polymer EDDY tip (VDW, Munich, Germany) with a 25.04 tip diameter and the Sonicmax sonic device (Maximum Dental Inc., Secaucus, NJ, USA) with one activation cycle. The EDDY (VDW) tip was placed in the canal 1 mm short of the working length and moved in a corono-apical direction at a frequency of 6 kHz and an amplitude of 5 mm for 1 minute to achieve MB activation. The MB (Merck KgaA) solution was renewed during the treatment.
  Interventions: Procedure: EDDY

INTERVENTIONS:
Procedure: Standard Needle Irrigation (SNI) — Standard Needle Irrigation (SNI):
  Utilizes standard needle irrigation techniques for activating the antimicrobial solution within the root canal.
  Arms: Standard Needle Irrigation (SNI) with MB Activation
Procedure: Passive Ultrasonic Irrigation (PUI — Passive Ultrasonic Irrigation (PUI):
  Employs ultrasonic energy to enhance the activation and effectiveness of the antimicrobial solution in the root canal.
  Arms: Passive Ultrasonic Irrigation (PUI) with MB Activation
Procedure: EndoActivator (EA) — EndoActivator (EA):
  Uses a sonic activation device to facilitate the distribution and activation of the antimicrobial solution in the root canal.
  Arms: EndoActivator(EA) with MB Activation
Procedure: EDDY — EDDY:
  Involves the use of a sonic activation device that operates at high frequency to activate the antimicrobial solution within the root canal.
  These descriptions focus on the general method and purpose of each intervention without delving into the specific procedural details already covered in the arm/group descriptions.
  Arms: EDDY with MB Activation

SUMMARY:
The decontamination of the root canal system from pathological microflora is essential for the success of endodontic treatment. Mechanical instrumentation and irrigation solutions, known as the chemomechanical process, are typically used for this purpose. However, due to the complex anatomy of teeth, residual microorganisms can remain, potentially affecting treatment success and weakening dentin walls. This has led to the development of more effective irrigation and disinfection systems.

Antimicrobial photodynamic therapy (aPDT) has emerged as a promising adjunct to traditional methods. aPDT is used to eliminate resistant microorganisms in various medical fields, including dentistry, and has been shown to effectively destroy oral bacteria in both planktonic and biofilm forms. However, aPDT is not a replacement for traditional endodontic procedures but can be used as an adjunct in root canal disinfection.

aPDT works through the presence of a photosensitizer, a radiation source with a sufficient wavelength, and oxygen, producing reactive oxygen species (ROS) that have a bactericidal effect. Methylene blue (MB) is a common photosensitizer, but it can cause tooth discoloration and is difficult to remove. Alternatives to MB are being sought.

Different activation techniques, such as passive ultrasonic irrigation (PUI) and sonic activation systems (SAS), have been developed to enhance the effectiveness of irrigation solutions. Studies have shown that PUI and SAS have similar effectiveness in traditional endodontic irrigation. Enterococcus faecalis is a particularly resistant bacterium involved in endodontic infections. While MB's effectiveness against E. faecalis is documented, there is a lack of studies comparing its effectiveness with ultrasonic and sonic systems in necrotic and periapical lesion teeth. There is also limited research on the discoloration potential and postoperative pain of MB when used with various activation systems. The study hypothesizes that there will be no significant difference in lesion healing, postoperative pain, and discoloration potential with different activation systems using aPDT.

DETAILED DESCRIPTION:
It is well known that the decontamination of the root canal system from pathological microflora is a prerequisite for the success of endodontic treatment. In addition to mechanical instrumentation, various irrigation solutions and intracanal medications are used to decontaminate the root canal from microorganisms. The combined use of mechanical instrumentation and irrigation solutions is referred to as the chemomechanical process. However, due to the complex anatomy of the tooth structure, such as lateral canals, isthmuses, dentinal tubules, and accessory canals, residual microorganisms may remain despite the completion of the chemomechanical process. This can negatively affect the success of the treatment. Additionally, it is noted that the dentin walls may weaken as a result of chemomechanical preparation. Therefore, researchers often emphasize the need for more effective irrigation and disinfection systems.

Recently, the application of antimicrobial photodynamic therapy (aPDT) has been shown to be a promising addition to traditional methods. Today, aPDT is used to eliminate resistant microorganisms in cancer treatment, macular degeneration, arterial plaque, arthritis treatment, and dentistry. aPDT has been reported to effectively destroy oral bacteria present in both planktonic and biofilm forms. However, researchers state that aPDT cannot replace traditional endodontic procedures but can be used as an adjunct in root canal disinfection.

The working principle of aPDT is based on the presence of a specific photosensitizer, a radiation source with a sufficient wavelength, and the presence of oxygen in the environment. As a result of the reaction caused by aPDT, reactive oxygen species (ROS) such as singlet oxygen and free radicals are produced, leading to a bactericidal effect. Thus, a wide range of microorganisms can be eliminated without encountering the resistance problem of current bacterial strains. Additionally, aPDT offers various advantages due to its repeatability, low toxicity, and minimally invasive approach.

Various photosensitizers and light sources with different wavelengths are available for use in aPDT. One of the most widely used photosensitizers in the literature is methylene blue (MB) from the phenothiazine salts group. However, it is known that MB is difficult to remove after application and can cause tooth discoloration. Therefore, alternative photosensitizers to MB are being sought. Today, the antimicrobial efficacy of MB is well recognized. Due to the low absorption exhibited by phenothiazine dyes, which are among the most commonly used photosensitizers, multiple applications are required for a high drug dose and effective treatment outcome. The effectiveness of solutions is not solely dependent on the properties of the solution but also varies with the method used. Although the traditional needle irrigation method (GII) is still in use, its effectiveness is limited. Another method, manual dynamic activation (MDA), involves creating a hydrodynamic force in the irrigation solutions by moving a gutta-percha that fits well into a shaped root canal in a corono-apical direction at the working length. This method is frequently used as it does not require additional materials.

With technological advancements, different methods have been developed to enhance the effectiveness of solutions. The passive ultrasonic irrigation (PUI) method shows effectiveness by causing acoustic streaming through the vibration it generates. The solution is activated during the application without any contact with the root canal walls. Another method, the sonic activation system (SAS), has been used in endodontics for years and has proven its effectiveness. Several SAS devices from different manufacturers have been developed. One commonly used device, Endoactivator, has a polymer tip and works through sinusoidal oscillation. Another widely used device, EDDY (VDW, Munich, Germany), oscillates at 5000-6000 Hz, causing three-dimensional movement in the root canal and triggering cavitation and acoustic streaming. Studies have shown that the effectiveness of PUI and SAS on traditional endodontic irrigation solutions is similar. Enterococcus faecalis (E. faecalis) is a gram-positive facultative bacterium. It is among the most resistant strains involved in the development of anaerobic and endodontic infections. Although detailed literature reviews have shown studies proving the effectiveness of MB on E. faecalis bacteria, there is no study comparing the effectiveness of MB solution in necrotic and periapical lesion teeth using ultrasonic and sonic systems. It has been found that there is no comprehensive study in the literature comparing the discoloration potential and postoperative pain of MB applied with various activation systems. The null hypothesis of the study is that there will be no significant difference in lesion healing, postoperative pain, and discoloration potential with different activation systems using aPDT.

ELIGIBILITY:
Inclusion Criteria:

* Teeth that had not undergone previous root canal treatment.
* Teeth with a single root and a single canal.
* Teeth with apical periodontitis.
* Teeth with periodontal lesion size less than 5 mm.
* Teeth without sinus tract or acute apical abscess.
* Patients without systemic diseases.
* Patients not pregnant.
* Patients who volunteered to participate in the study.
* Patients who agreed to attend follow-up sessions.

Exclusion Criteria:

* Patients using medications such as antihypertensives or antidiabetics that could affect root canal treatment outcomes.
* Patients using corticosteroids or antibiotics.
* Patients with acute pain or extraoral swelling.
* Patients with a history of sinus tract or acute apical abscess.
* Patients with systemic diseases.
* Patients who are pregnant.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-07-14 (Actual)

PRIMARY OUTCOMES:
Reduction in Bacterial Load | Up to 6 months
  This study aims to evaluate the effectiveness of antimicrobial photodynamic therapy (aPDT) using different irrigation activation techniques in teeth with apical periodontitis. The study will be conducted as a randomized, parallel-group clinical trial with four intervention groups: Standard Needle Irrigation (SNI), Passive Ultrasonic Irrigation (PUI), EndoActivator (EA), and EDDY.

CONTACTS AND LOCATIONS:
Overall Officials: Özge Hür Şahin, DDS, Study Director — University of Health Sciences Gülhane; Zeliha Uğur Aydın, Assoc. Prof., Study Chair — University of Health Sciences Gülhane
Locations (1):
- University of Health Sciences Gulhane, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We are currently undecided about sharing individual participant data (IPD) with other researchers. A decision will be made based on further discussions within the research team, ethical considerations, and the potential value of the data for future research. We will update this section once a final decision has been reached.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From baseline to 6 months post-treatment
Access Criteria: undecided

REFERENCES:
- [Result] Asnaashari M, Mojahedi SM, Asadi Z, Azari-Marhabi S, Maleki A. A comparison of the antibacterial activity of the two methods of photodynamic therapy (using diode laser 810 nm and LED lamp 630 nm) against Enterococcus faecalis in extracted human anterior teeth. Photodiagnosis Photodyn Ther. 2016 Mar;13:233-237. doi: 10.1016/j.pdpdt.2015.07.171. Epub 2015 Aug 1. PMID 26241781
- [Result] Er Karaoglu G, Ugur Ydin Z, Erdonmez D, Gol C, Durmus M. Efficacy of antimicrobial photodynamic therapy administered using methylene blue, toluidine blue and tetra 2-mercaptopyridine substituted zinc phthalocyanine in root canals contaminated with Enterococcusaecalis. Photodiagnosis Photodyn Ther. 2020 Dec;32:102038. doi: 10.1016/j.pdpdt.2020.102038. Epub 2020 Oct 1. PMID 33010484
- [Result] da Silva CC, Chaves Junior SP, Pereira GLD, Fontes KBFDC, Antunes LAA, Povoa HCC, Antunes LS, Iorio NLPP. Antimicrobial Photodynamic Therapy Associated with Conventional Endodontic Treatment: A Clinical and Molecular Microbiological Study. Photochem Photobiol. 2018 Mar;94(2):351-356. doi: 10.1111/php.12869. Epub 2018 Jan 19. PMID 29166538